CLINICAL TRIAL: NCT06226545
Title: A Phase 2, Proof-of-Concept, Randomized, Double-Masked, Placebo-Controlled Study to Determine the Efficacy and Safety of LASN01 in Patients With Thyroid Eye Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of LASN01 in Patients With Thyroid Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lassen Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LASN01-CL-2201
Record Dates: First submitted 2023-12-14; First posted 2024-01-26 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Thyroid Eye Disease; Graves Ophthalmopathy; Graves Orbitopathy; Thyroid Associated Ophthalmopathy; Endocrine System Diseases; Orbital Diseases; Proptosis; Eye Diseases
MeSH Terms: conditions — Graves Ophthalmopathy; Endocrine System Diseases; Orbital Diseases; Exophthalmos; Eye Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double masked treatment arms for patients without prior anti-IGF-1R treatment, and open-label treatment arm for patients with prior teprotumumab treatment
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Randomized low-dose LASN01 (anti-IGF-1R-naïve TED) (Experimental)
  Interventions: Drug: LASN01
- Randomized high-dose LASN01 (anti-IGF-1R-naïve TED) (Experimental)
  Interventions: Drug: LASN01
- Randomized placebo (anti-IGF-1R-naïve TED) (Placebo Comparator)
  Interventions: Drug: Placebo
- Open-label high dose LASN01 (post-teprotumumab, US only) (Experimental)
  Interventions: Drug: LASN01

INTERVENTIONS:
Drug: LASN01 — Low dose of LASN01 will be administered intravenously.
  Other Names: Low-dose LASN01
  Arms: Randomized low-dose LASN01 (anti-IGF-1R-naïve TED)
Drug: LASN01 — High dose of LASN01 will be administered intravenously.
  Other Names: High-dose LASN01
  Arms: Randomized high-dose LASN01 (anti-IGF-1R-naïve TED)
Drug: Placebo — Placebo will be administered intravenously.
  Other Names: Placebo to match
  Arms: Randomized placebo (anti-IGF-1R-naïve TED)
Drug: LASN01 — High dose of LASN01 will be administered intravenously.
  Other Names: High-dose LASN01
  Arms: Open-label high dose LASN01 (post-teprotumumab, US only)

SUMMARY:
LASN01 is a novel, fully human antibody directed against the human IL-11 receptor being developed for treatment of patients with thyroid eye disease (TED).

The primary and secondary objectives of this study are to evaluate the safety, treatment effect, and pharmacokinetics of LASN01 administered IV in patients with TED with no prior anti-IGF-1R treatment or in patients with TED who have previously received teprotumumab treatment.

DETAILED DESCRIPTION:
This clinical trial (LASN01-CL-2201) comprises a multiple-dose design in 3 parallel treatment arms for patients with TED with no prior anti-IGF-1R treatment, and a 4th treatment arm for patients with TED who have previously received teprotumumab treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years of age at the time of Screening
2. Clinical diagnosis of Graves' disease associated with active TED
3. Moderate-to-severe active TED
4. Female patients must be nonpregnant, nonlactating, surgically sterile for ≥6 months, or agree to use a highly effective method of contraception. Males must be surgically sterile or agree to use a highly effective method of contraception.
5. No previous:

   1. Medical treatment for TED, with the exception of:

      * Local supportive measures;
      * Mycophenolate, and oral or injectable steroids;
      * Immunomodulating therapies
      * For the open-label treatment arm only: Previous treatment with teprotumumab is required.
   2. Orbital surgery
   3. Orbital radiation
6. Patients

   * Without prior anti-IGF-1R treatment: less than 15 months from onset of TED symptoms
   * With prior teprotumumab treatment: depending on time of diagnosis or reactivation of disease

Exclusion Criteria:

1. Patients with 2 mm proptosis decrease between Screening and Day 1, or a 1-point decrease on the CAS 7-point scale between Screening and Day 1
2. Patients with a known decreased best corrected visual acuity due to optic neuropathy as defined by a decrease in vision of 3 lines on the Snellen chart, new visual field defect, or color defect secondary to optic nerve involvement within the last 6 months before Screening; or any known optic neuropathy or compression or any neurologic or neuro-ophthalmologic condition that may result in visual field loss.
3. Previous or any planned orbital irradiation/radiotherapy or orbital surgery for TED during the study period (ie, treatment and FU)
4. Use of oral and/or IV corticosteroid for conditions other than TED in the 6 weeks before Day 1 (topical steroids for conditions other than TED are allowed)
5. Active autoimmune disorder(s) requiring or likely to require treatment (other than Grave's disease and TED) that would interfere with study assessments, as determined by the PI or designee
6. Any previous use of anti-IGF-1R monoclonal antibody (eg, teprotumumab) at any time, with exception to the open-label post-teprotumumab treatment arm where prior use of teprotumumab is required
7. Use of selenium within 3 weeks before Day 1 or expected use during the clinical trial (multivitamins that include selenium are allowed in usual doses)
8. Use or expected use of biotin (including multivitamins that include biotin) within 2 days before any laboratory collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Changes in proptosis in the study eye compared to baseline as assessed by Exophthalmometer | Day 1-Day 253
For randomized treatment arms: Number of participants with adverse events receiving LASN01 compared to placebo | Day 1-Day 253
For open-label treatment arm: Number of participants with adverse events receiving LASN01 | Day 1-Day 253

SECONDARY OUTCOMES:
Change in Clinical Activity Score (CAS) in the study eye compared to baseline as assessed by CAS evaluation | Day 1-Day 505
Change in lid aperture in the study eye compared to baseline as measured by the changes of the distance between the lid margins | Day 1-Day 505
Change in lid retraction in the study eye compared to baseline as assessed by measurement of margin reflex distance 1 and 2 | Day 1-Day 505
Change in lagophthalmos in the study eye compared to baseline as assessed by presence or absence of lagophthalmos | Day 1-Day 505
Change in Von Graefe's sign in the study eye compared to baseline as assessed by presence or absence of Von Graefe's sign | Day 1-Day 505
Change in extraocular movements in the study eye compared to baseline as assessed by duction testing | Day 1-Day 505
Change in diplopia in the study eye compared to baseline as assessed by Bahn-Gorman Scale | Day 1-Day 505

CONTACTS AND LOCATIONS:
Locations (15):
- United States (10):
  - Site 111, Beverly Hills, California
  - Site 105, Palo Alto, California
  - Site 101, San Diego, California
  - Site 103, Miami, Florida
  - Site 108, Livonia, Michigan
  - Site 112, Las Vegas, Nevada
  - Site 110, Wilmington, North Carolina
  - Site 106, Houston, Texas
  - Site 104, Houston, Texas
  - Site 109, Seattle, Washington
- Spain (2):
  - Site 302, Córdoba
  - Site 301, Seville
- United Kingdom (3):
  - Site 201, London
  - Site 206, London
  - Site 204, Newcastle upon Tyne